CLINICAL TRIAL: NCT07003126
Title: A Cohort Study on Treating Primary Nocturnal Enuresis by Regulating Central-Peripheral Circadian Rhythm
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-PWDL-13
Record Dates: First submitted 2025-05-25; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Primary Nocturnal Enuresis
Keywords: Primary Nocturnal Enuresis; Circadian Rhythm; Treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Circadian Rhythm Intervention Combined with Bladder Training (Experimental): The study population consists of children diagnosed with primary nocturnal enuresis according to the diagnostic criteria established by the International Children's Continence Society (ICCS). Participants will receive bladder training including fluid intake modification, micturition desire-relaxation training and sphincter control training combined with circadian rhythm interventions, including sleep hygiene education, chronotype-guided bedtime scheduling, and morning bright light therapy. Clinical symptom severity and key pathophysiological measures will be assessed at baseline and 6 months after intervention initiation.
  Interventions: Behavioral: Circadian Rhythm Intervention Combined with Bladder Training
- Bladder Training (basic treatment for enuresis) (Active Comparator): The study population consists of children diagnosed with primary nocturnal enuresis according to the ICCS criteria. Participants will undergo bladder training interventions, specifically including fluid intake modification, micturition desire-relaxation training and sphincter control training. The clinical symptom progression will be monitored, and key outcome measures will be prospectively collected at two timepoints: baseline (pre-intervention) and 6 months after intervention initiation.
  Interventions: Behavioral: Bladder Training (basic treatment for enuresis)

INTERVENTIONS:
Behavioral: Circadian Rhythm Intervention Combined with Bladder Training — Participants diagnosed with primary nocturnal enuresis will be screened at Shanghai Children's Medical Center, and eligible patients will be enrolled. Participants will be randomly assigned to the Bladder Training Combined with Circadian Rhythm Intervention Group, which will receive a 6-month integrated protocol encompassing bladder training and circadian rhythm intervention. The bladder training component includes fluid intake restriction, micturition desire-relaxation training, and sphincter control training. Circadian rhythm interventions involve sleep hygiene education, chronotype-guided bedtime scheduling, and morning bright light therapy.
  Arms: Circadian Rhythm Intervention Combined with Bladder Training
Behavioral: Bladder Training (basic treatment for enuresis) — Participants diagnosed with primary nocturnal enuresis will be screened at Shanghai Children's Medical Center, and those meeting eligibility criteria will be enrolled. Participants will be randomized to the Bladder Training Only Group, which will receive a 6-month intervention comprising fluid intake restriction, micturition desire-relaxation training, and sphincter control training.
  Arms: Bladder Training (basic treatment for enuresis)

SUMMARY:
Primary nocturnal enuresis (PNE), a prevalent pediatric disorder, suffers from therapeutic limitations characterized by low efficacy and high relapse rates. Targeting its core pathophysiology could significantly improve treatment outcomes. Growing evidence implicates circadian dysregulation in PNE pathogenesis. Our preliminary fMRI cohort identified abnormal functional connectivity between the suprachiasmatic nucleus (SCN, the central circadian pacemaker) and superior temporal gyrus in PNE patients, with clinical data confirming circadian realignment correlates with symptom remission. Small-scale pilot studies and clinical observations indicate that modulating central and peripheral circadian rhythms significantly alleviates PNE symptoms. This study will establish a circadian-focused PNE cohort to quantify therapeutic efficacy and elucidate underlying mechanisms, ultimately driving the development of mechanism-based therapies for PNE.

DETAILED DESCRIPTION:
The intervention training will last for 6 months. Researchers will compare the therapeutic efficacy of the "Circadian Rhythm Intervention Combined with Bladder Training Group (treatment group)" and the "Bladder Training (basic treatment for enuresis) Only Group (control group)" for PNE.

Participants will be assigned to either the "Circadian Rhythm Intervention Combined with Bladder Training Group (treatment group)" or "Bladder Training (basic treatment for enuresis) Only Group (control group)" through stratified block randomization matching participants by sex (male/female), age (in years), and enuresis frequency. Within each stratified subgroup, block randomization with a 1:1 allocation ratio will be implemented using computer-generated random sequences, ensuring balanced demographic distribution between the two intervention arms while maintaining concealment of allocation sequence.

In the "Circadian Rhythm Intervention Combined with Bladder Training Group (treatment group)", participants will receive a 6-month behavioral therapy including both bladder training and circadian rhythm intervention. Bladder training combined with circadian rhythm interventions involves sleep hygiene optimization, individualized chronotype alignment, morning bright light therapy and bladder training component. The bladder training component (basic treatment for enuresis) includes fluid intake modification, micturition desire-relaxation training, and sphincter control training. Clinical symptom severity and key pathophysiological parameters will be evaluated at baseline and at 6 months post-intervention.

In the "Bladder Training Only Group (control group)", participants will receive a 6-month behavioral therapy including only bladder training. The bladder training component (basic treatment for enuresis) includes fluid intake modification, micturition desire-relaxation training, and sphincter control training. Clinical symptom severity and key pathophysiological parameters will be evaluated at baseline and 6 months post-intervention.

The investigators will compare changes in enuresis improvement rate, resting-state functional magnetic resonance imaging data, sleep physiological parameters, salivary melatonin levels, diurnal and nocturnal urine volume, standardized bladder capacity, and grade scoring of the micturition desire-awakening function before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis according to the ICCS criteria:

   At least one episode of involuntary nighttime urination per month for more than 3 months.

   No abnormalities in routine urinalysis. No period of bedwetting-free days lasting more than 6 months, except for organic diseases.
2. Age: 5 to 15 years (inclusive), regardless of gender.
3. Right-handedness (as assessed by the Annett Hand Preference Questionnaire)

Exclusion Criteria:

1. Secondary nocturnal enuresis;
2. History of head trauma, neurological disorders, psychosurgery, or major physical conditions (including autism spectrum disorder, epilepsy, cerebral palsy);
3. Contraindications to fMRI.
4. Note: Mild comorbidities commonly associated with primary nocturnal enuresis (e.g., ADHD) are permitted but must be included as covariates in statistical analyses.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Enuresis Improvement Rate | From enrollment to the end of treatment at 6 months
  The enuresis improvement rate is the sum of the complete and partial response rates.
  No response: <50% reduction. Partial response: 50 to 99% reduction. Complete response: 100% reduction.

SECONDARY OUTCOMES:
Resting-State Functional Magnetic Resonance Imaging (fMRI) Data | From enrollment to the end of treatment at 6 months
  Resting-state fMRI data will be acquired to characterize brain functional networks, with a focus on analyzing functional connectivity between the suprachiasmatic nucleus and superior temporal gyrus.
Diurnal and Nocturnal Urine Volume | From enrollment to the end of treatment at 6 months
  Participants will complete at least one 24-hour fluid intake and voiding diary per week, including diurnal and nocturnal urine volume recorded pre-treatment, during treatment, and post-treatment.
  Daytime voiding will be measured using graduated plastic cylinders for each urination. Nocturnal voiding will be recorded by wearing pre-weighed diapers (with urine volume calculated by weighing the diapers the next day) or through timed voiding upon waking during the night.
  The average total diurnal and nocturnal urine volume during each recorded period will be calculated as the participant's diurnal and nocturnal urine volume at different time points.
Heart Rate Variability | From enrollment to the end of treatment at 6 months
  Continuous measurement of beat-to-beat intervals assessed via research-grade wearable actigraphy, using artificial intelligence-driven chronobiological analytics to extract features.
  Unit of Measure: Milliseconds
Polysomnography-Validated Sleep Metrics | From enrollment to the end of treatment at 6 months
  Sleep efficiency validated against polysomnography benchmarks and derived from wearable actigraphy data streams.
  Unit of Measure: Percent (%)
Grade scoring of the micturition desire-awakening function | From enrollment to the end of treatment at 6 months
  The grade scoring of the micturition desire-awakening function based on the average awakening ability each night. The grade scoring of the micturition desire-awakening function is as follows:
  Grade 5: Remains asleep most of the time after urination. Grade 4: Only awakens after completely wetting the bed. Grade 3: Awakens only after urinating a significant amount and then goes to the toilet to void the remaining urine.
  Grade 2: Awakens after urinating a small amount and then goes to the toilet to void the remaining urine.
  Grade 1: Awakened by the urge to urinate, without wetting the bed.
Standardized Bladder Capacity | From enrollment to the end of treatment at 6 months
  Standardized bladder capacity = bladder capacity/body surface area. Compare the standardized mean bladder capacity as well as the maximum and minimum daytime/nighttime bladder capacity changes from baseline to 6 months.
  The term mean daytime bladder capacity refers to the average volume of voided urine measured on the frequency volume chart throughout a 24-hour cycle.
  The term maximum/minimum daytime bladder capacity refers to the largest/smallest volume of voided urine measured on the frequency volume chart during the day. It excludes the first morning void.
  The term maximum/minimum nighttime bladder capacity refers to the largest/smallest volume of voided urine measured on the frequency volume chart during the night. It includes the first morning void.
Salivary Melatonin Levels | From enrollment to the end of treatment at 6 months
  Saliva samples (2 mL each) will be collected from children with PNE at 4-hour intervals starting at 09:00, yielding seven timepoints (09:00, 13:00, 17:00, 21:00, 01:00, 05:00, and 09:00 the following day) within a ±1-hour window. Collections at 21:00, 01:00, and 05:00 will be performed under dim-light conditions (ambient illumination <30 lux).
  Salivary melatonin concentrations will be quantified using liquid chromatography-tandem mass spectrometry-a rapid, sensitive, and reliable method validated for low-abundance hormone detection in saliva.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai children's medical center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Austin PF, Bauer SB, Bower W, Chase J, Franco I, Hoebeke P, Rittig S, Vande Walle J, von Gontard A, Wright A, Yang SS, Neveus T. The standardization of terminology of lower urinary tract function in children and adolescents: update report from the Standardization Committee of the International Children's Continence Society. J Urol. 2014 Jun;191(6):1863-1865.e13. doi: 10.1016/j.juro.2014.01.110. Epub 2014 Feb 4. PMID 24508614